CLINICAL TRIAL: NCT00673023
Title: Study the Role of Polymorphism at the CETP Gene Locuse in the Determining Lipid Profile Response to Dietary Change
Brief Title: Study the Role of Genetic Variation in the Determining Lipid Profile Response to Dietary Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tabriz University (Other)
Responsible Party: vice-chancellor for reseach, Tabriz University, Deputy of Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 8641
Record Dates: First submitted 2008-05-04; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Other: Dietary experiments
- 2 (Experimental)
  Interventions: Other: Dietary experiments
- 3 (Experimental)
  Interventions: Other: Dietary experiments

INTERVENTIONS:
Other: Dietary experiments — Dietary Supplement: high PUFA diet followed by high SFA diet

SUMMARY:
The purpose of this study is to determine whether plasma lipoproteins and lipid responsiveness to a dietary modification is influenced by CETP gene polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers

Exclusion Criteria:

* History of any cardiovascular diseases
* type 1 diabetes
* type 2 diabetes
* use of lipid-lowering medications
* hypertension
* pregnancy
* Current intake of vitamins and supplements
* History of endocrin disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Noori, PhD, Study Director — Tabriz University